CLINICAL TRIAL: NCT04740424
Title: A Phase 1, Open-Label, First-in-Human Study to Evaluate the Safety and Anti-tumour Activity of FS222, a CD137/PD-L1 Bispecific Antibody, in Subjects With Advanced Malignancies
Brief Title: FS222 First in Human Study in Patients With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: invoX Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FS222-19101
Record Dates: First submitted 2021-01-28; First posted 2021-02-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: Immuno-oncology; bispecific antibody; dose escalation; cohort expansion; CD137; PD-L1; F-star; 4-1BB; Immunotherapy
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FS222 Q4W (Experimental): The initial cohorts will enroll sequentially as single participant cohorts. If no DLT or ≥Grade 2 study drug related adverse event is observed, then dosing will proceed in a 3+3 design. Additional participants will be recruited into the PK/PD expansion cohorts at dose levels deemed safe during dose escalation. Once a tolerated dose has been established participants will be recruited into tumour-specific expansion cohorts.
  Interventions: Drug: FS222

INTERVENTIONS:
Drug: FS222 — Dosing of participants will occur intravenously (IV), at a fixed dose in treatment cycles once every 4 weeks (Q4W) until disease progression or unacceptable toxicity.

SUMMARY:
This study will be conducted in adult participants diagnosed with advanced tumours to characterize the safety, tolerability, pharmacokinetics (PK), and activity of FS222. This is a Phase 1, multi-center, open label, multiple-dose, first in human study, designed to systematically assess safety and tolerability, and to identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) for FS222 in participants with advanced tumours. Pharmacokinetics, pharmacodynamics, immunogenicity, and response will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Participants with histologically or cytologically confirmed, locally advanced, unresectable or metastatic solid tumours for whom standard therapy has proven to be ineffective, intolerable or is considered inappropriate. This criterion does not apply to the PK/PD expansion cohort, where tumour-specific criteria will apply instead.
* No more than 1 line of prior therapy with ICB treatment. Exceptions as defined in protocol for PK/PD expansion cohorts will apply.
* Participants who have received prior ICB, or any concurrent chemotherapy, radiotherapy, investigational, biologic or hormonal therapy for cancer treatment may be eligible for enrolment following a washout period.
* Participants who have received prior anti-PD-L1 therapy are eligible if PD-L1 therapy was discontinued ≥6 months prior to entry into the study.
* Participants who have failed a prior ICB regimen should document it.
* Measurable disease. Exceptions as defined in protocol for PK/PD expansion cohorts will apply.
* Eastern Cooperative Oncology Group Performance Status ≤1.
* The participant agrees to undergo a mandatory pre-treatment and on-treatment biopsy of the tumour. Certain exceptions apply.
* Highly effective contraception.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Participants with clinically relevant COVID-19 disease risk will be excluded from enrolment during the COVID-19 pandemic.
* Concurrent enrolment in another clinical study with the exception of non-interventional/observational studies or the follow-up period of an interventional study.
* Prior treatment with CD137 agonist mAb or other experimental agonists.
* For participants who have received prior ICB, participants must not have received more than 1 line of prior treatment with ICB(s). Exceptions as defined in protocol for PK/PD expansion cohorts will apply.
* Participants with active autoimmune disease.
* Receipt of any live virus vaccine within 30 days prior to the first dose of study drug.
* Receipt of a live attenuated vaccine within 30 days prior to the first dose of study drug.
* History of uncontrolled intercurrent illness.
* Psychological, familial, sociological or geographical conditions that do not permit compliance with the protocol.
* Judgment by the investigator that the participant is unsuitable to participate in the study, and the participant is unlikely to comply with study procedures, restrictions and requirements.
* Significant laboratory abnormalities.
* Known infections.
* Uncontrolled CNS metastases, primary CNS tumours with CNS metastases as only measurable disease. Exceptions as defined in protocol for PK/PD expansion cohorts will apply.
* Prior history of any Grade ≥3 irAE that has not improved to Grade ≤1, except for endocrine deficiencies that are managed by HRT; significant treatment-related cytokine release syndrome; systemic inflammatory response syndrome.
* Current use of immunosuppressive agents, prior organ transplantation requiring immunosuppression, hypersensitivity or intolerance to mAb or their excipients, or persisting toxicity related to prior therapy of Grade >1 NCI CTCAE Version 5.0 .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Presence of adverse events (AEs) and serious adverse events (SAEs) | 15 months
  Safety and tolerability will be evaluated by collection of AEs and SAEs according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.
Determination of a maximum tolerated dose (MTD) by evaluation of DLTs | 28 days
  Toxicity will be evaluated according to the NCI CTCAE Version 5.0.
Determination of a recommended Phase 2 dose (RP2D) by evaluation of DLTs | 28 days
  Toxicity will be evaluated according to the NCI CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (21):
- Australia (2):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - One Clinical Research Perth, Perth, Western Australia
- Arensia Exploratory Medicine, LLC, Tbilisi, Georgia
- SLK Kliniken Heilbronn GmbH, Heilbronn, Baden-Wurttemberg, Germany
- Radboud Universitair Medisch Centrum, Nijmegen, Gelderland, Netherlands
- Poland (2):
  - Centrum Medyczne Poznan - PRATIA - PPDS, Poznan, Greater Poland Voivodeship
  - MCM Krakow - PRATIA - PPDS, Krakow
- Romania (2):
  - Prof. Dr. Alexandru Trestioreanu Oncologic Institute, Bucharest
  - Prof Dr I Chiricuta Institute of Oncology, Cluj-Napoca
- Spain (12):
  - Clinica Universidad Navarra, Pamplona, Navarre
  - NEXT - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala d'Oncologia de Badalona, Barcelona
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria
  - Instituto de Investigación Sanitaria Fundación Jimenez Díaz, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - NEXT - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Universitary Hospital Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided